CLINICAL TRIAL: NCT06174948
Title: The Use of the CUE1/CUE1+ Device in People With Idiopathic Parkinson's Disease and Related Disorders: A Feasibility Study
Brief Title: The Use of the CUE1/CUE1+ in People With Parkinson's Disease and Related Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other); Homerton University Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 333484
Record Dates: First submitted 2023-11-30; First posted 2023-12-18 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease and Parkinsonism; Progressive Supranuclear Palsy; Different Types of Tremor Including Essential Tremor; Dystonia; Multiple System Atrophy; Corticobasal Degeneration; Vascular Parkinsonism; Orthostatic Tremor
Keywords: CUE1, Parkinson's disease, movement disorders
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Supranuclear Palsy, Progressive; Dystonia; Multiple System Atrophy; Corticobasal Degeneration; Movement Disorders

STUDY DESIGN:
Intervention Model Description: Initially, 10 people with idiopathic Parkinson's disease and 10-20 people with related movement disorders are firstly assigned into a single group study to investigate the feasibility, safety and tolerability of the CUE1 device.
  Then a subgroup of participants (e.g., 30-40 new participants) with idiopathic Parkinson's disease only will be randomly allocated to one of the two intervention Groups; one group will receive the CUE1+ intervention at loud settings while the other at silent settings. The outcome assessor and statistician the group of the participants. Participants will know in which group they are but they do not know which is the active and which the passive intervention. This intervention is the main of this study and is double blind.
Who Masked: Participant, Outcomes Assessor
Masking Description: The masking only applies to investigation for a subgroup of people with Parkinson's disease (e.g., 30-40 participants) There is no masking for the single group intervention of people with Parkinson's related disorders and the first 10 participants with Parkinson's disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- people with Parkinson's disease and related disorders (Experimental): Intervention
  All participants with Parkinson's related disorders and the first 10 participants with Parkinson's will use the CUE1 device as follows:
  * 1-2/9 weeks in the study: once a day for a continuous duration of 2 hours in the morning, 1 hour after taking the medication (if any) for PD or related disorder, every single day;
  * 4-5/9 weeks in the study: once a day for a continuous duration of 8 hours, starting from morning, 1 hour after taking the medication (if any) for PD or related disorder, every single day;
  * 7-8/9 weeks in the study: only at night, through all night, every single night and not during the day at all;
  15-20 participants with Parkinson's disease will use the CUE1+ device at loud settings for 12 continuous weeks, as above the participants during weeks 4-5.
  Interventions: Device: CUE1 non-invasive device; Device: CUE1+ device active vs sham CUE1+ device
- People with Parkinson's disease (Sham Comparator): 15-20 participants with Parkinson's disease will use the CUE1+ device sat silent settings for 12 continuous weeks, as above the participants during weeks 4-5 and compared to the active CUE1+ intervention with people with Parkinson's disease only as above
  Interventions: Device: CUE1+ device active vs sham CUE1+ device

INTERVENTIONS:
Device: CUE1 non-invasive device — This is a 9-week feasibility study which will involve wearing the CUE1 device on a daily basis at participants' homes while they continue their usual activities of daily living (ADL). The CUE1 is a non-invasive medical device which delivers low frequency metronomes like tactile cueing and high frequency focused vibrotactile stimulation. All participants will be using the same pre-programmed settings for the CUE1 device which are: vibration strength delivered at 80%, pulse length 800 milliseconds (ms), and rest length 800ms as set at baseline and will not change. The CUE1 device is attached to the skin via an adhesive patch which has been dermatologically tested and approved. Participants will be provided with the adhesive patches and shown how to use them and the CUE1 device by the research team.
  Arms: people with Parkinson's disease and related disorders
Device: CUE1+ device active vs sham CUE1+ device — 30-40 participants with idiopathic Parkinson's disease only will be randomly allocated to one of two interventions groups: one group will use the active CUE1+ device while the other group will use the CUE1+ at silent settings (e.g., sham device). All participants will use their device in the same way which is starting the usage from the morning, within an hour once they took their medications for Parkinson's (if any) and continue using the device for 8 hours, once a day, every day for 12 weeks
  Other Names: CUE1+ device sham

SUMMARY:
People with Parkinson's disease (PD) commonly experience a range of both motor (e.g., bradykinesia, rigidity, tremor, and postural instability) and non-motor (e.g., fatigue, psychiatric and behavioural disturbances, autonomic dysfunction, cognitive impairment, sleep dysfunction and olfactory loss) features. Currently, it is challenging to alleviate these symptoms with first-line treatment, the medications such as levodopa. The CUE1 is a non-invasive device, which is approved for sale in the UK market as a Class I low risk device. It is worn on the sternum or other part of the body such as the forearm and attaches to the skin via an adhesive patch which has been dermatologically tested and approved.

The CUE1 delivers pulsing cueing and vibrotactile stimulation to help improve symptoms in people with PD and it has shown to be effective in doing so in previous small case studies. This 9-week feasibility study aims to investigate the feasibility, safety, tolerability and effect of using the CUE1 as an intervention to improve motor and non-motor symptoms in people with PD and related movement disorders. People with clinical diagnosis of idiopathic PD and related disorders including those with progressive supranuclear palsy, multiple system atrophy, corticobasal degeneration, orthostatic tremor and vascular Parkinsonism as well as atypical dystonias and tremor disorders aged over 18 years old who have the capacity to provide a written consent form to take part in the study, will receive as intervention to wear the CUE1 device at home, on daily basis while carrying out their activities of daily living. Participants will also have to attend face-to-face appointments of approximately half a day, to discuss how they are getting on with using the CUE1 and complete questionnaires on their symptoms, walking, balance, and movement tests as well as a participant's clinical diary.

DETAILED DESCRIPTION:
Parkinson's disease (PD) may be the fastest growing neurodegenerative disease in the world (Bloem et al., 2021). Pathologically, it is characterised by the loss of the dopaminergic neurons within the substantia nigra pars compacta (SNc) and other pigmented nuclei of the brainstem. At present, the cost of healthcare for the estimated 145,000 people living with PD in the United Kingdom is over £728 million per year rising to a total economic impact of £3.6 billion (Weir et al. 2018). If current projections are correct of people with PD, this will double by 2040 (Dorsey et al. 2018), consequently the figure may exceed £7.2 billion. Most people affected are 60 years or above. However, there are many people who are diagnosed at a younger age. Common clinical manifestations of PD include a range of both motor (e.g., bradykinesia, rigidity, tremor, and postural instability) and non-motor (e.g., fatigue, psychiatric and behavioural disturbances, autonomic dysfunction, cognitive impairment, sleep dysfunction and olfactory loss) features.

The motor features can be present anywhere in the body. Some of the common features are lack of facial expression, low volume speech, stiffness and slowness of movements. Further, gait and balance are often affected. People with PD tend to have a festinating gait, and/or experience postural instability with or without freezing of gait (FOG) which may occur when initiating walking, standing from sitting, turning, and passing through narrow passages or certain circumstances such as approaching a destination (Nutt et al., 2011) or dual tasking (DT) (Bloem et al., 2000; Jacobs et al., 2014; Isaacson et al., 2018). Postural instability, gait problems and FOG may significantly affect a person's ability to perform ADL, increase their falls risk (Muslimovic et al., 2008; Lamont et al., 2017) and reduce their quality of life (QoL). Approximately 70% of people with PD will fall in a year period which can often result in serious consequences including injuries (e.g., fractures and traumatic brain injury) which further increase morbidity, mortality, and healthcare and personal costs (Farombi et al., 2016).

Currently, there is no cure for PD or treatment options available that can slow down the progression of this condition. However, all people with PD are provided options to treat the signs and symptoms of the condition to support their ability to participate in ADL that are meaningful to them (Huber et al., 2011). First line therapy, the dopaminergic medications, have some impact on motor symptoms in PD but rarely get people back to a "normal" state (Killane et al., 2015). People often remain significantly limited in their ADL during 'OFF' state but even during 'ON' state, many features of PD do not respond adequately despite optimal pharmacotherapy (Shukla et al., 2012). Moreover, the usage of medication often has serious side effects, particularly in older adults. The average person living with PD may be taking nine doses of medication a day (Grosset et al., 2007). Thus, drug resistance is another concern and dose limiting side effects is a barrier to successful deployment of pharmacotherapy (Killane et al., 2015). This issue increases with disease progression because neurodegeneration progressively involves non-dopaminergic brain areas. As a result, various non-pharmacological, non-invasive interventions have been developed to manage sensory dysfunction, a major problem in people with PD, associated with PD symptoms (Conte et al., 2013). Cueing and vibrotactile sensory stimulation are two such examples that have been used to modulate sensory dysfunction in people with PD, especially the sensorimotor integration problems.

Cueing is a mechanism of applying an external temporal or spatial stimulus to facilitate movement initiation and continuation and it can be somatosensory, auditory, attentional or visual (Nieuwboer et al., 2007; Muthukrishnan et al., 2019). It is reported to work by shifting habitual motor control to goal directed motor control (Redgrave et al., 2010). Many studies have demonstrated that cueing helps to improve postural control, balance, FOG (van Wegen et al., 2006; Nieuwboer et al., 2007; Munoz-Hellin et al., 2013; Spaulding et al., 2013; Muthukrishnan et al., 2019), as well as DT performance in activities involving the upper (Heremans et al., 2016; Park & Kim, 2021) and lower (Rochester et al., 2007; 2009; 2010 (a); 2010(b); Fok et al., 2010; Mak et al., 2013; Beck et al., 2015; Chomiak et al., 2017; Mancini et al., 2018; Stuart & Mancini, 2020) limbs in people with PD. However, many cueing modalities used for the research purposes in the laboratory environments cannot be easily replicated in people's homes. Thus, a recent narrative review recommends the development of cueing wearable systems that can be used at home or in the community to improve gait and posture in PD (Muthukrishnan et al., 2019).

Interventions utilising vibrotactile sensory stimulation in PD can be split into two main groups: a) whole body vibrotactile stimulation and b) focused (e.g., targeted) vibrotactile stimulation. The results on the effectiveness of whole body vibrotactile stimulation on sensory dysfunction and motor symptoms are mixed with a large variation being reported from none to small improvement on motor symptoms, balance, gait and mobility (Dincher et al., 2019). On the other side, focused vibrotactile stimulation which is a non-invasive neuromodulation technique used by somatosensory cues (e.g., tactile/somatosensory cueing) to apply gentle vibrations to focal joints in the body may have a more positive and consistent effect (Basta et al., 2011; Pfeifer et al., 2021). Trials which include cylindrical vibration devices on the triceps (Pereira et al., 2016), a vibrotactile waistband around the abdomen in FOG (Goncalves et al., 2018), vibrotactile insoles to reduce falls (Otis et al., 2016) and a proprioceptive stabiliser on postural instability (Volpe et al., 2014) show promising results. The CUE1 is a non-invasive medical device which utilises a metronome-like pulsed vibration which represents both auditory and somatosensory low frequency cueing and high frequency focused vibrotactile stimulation to help improve motor task performance in people with PD (Tan et al., 2021; Ong et al., 2022; Wilhelm et al., 2022). It is a CE marked and an MHRA registered non-invasive medical device.

Like other cueing and vibrotactile stimulation devices, the CUE1 stands out as a non-invasive medical instrument. It employs a metronome-like pulsed vibration, incorporating both auditory and somatosensory low-frequency cueing, along with high-frequency targeted vibrotactile stimulation. This design aims to enhance motor task performance in individuals with PD (Tan et al., 2021; Ong et al., 2022; Wilhelm et al., 2022). Preliminary assessments of employing the CUE1 indicated an overall enhancement of 16.75% in motor symptoms, as evidenced in the White Paper on Proof of Concept from 2019. This improvement was observed not only in the MDS-UPDRS Part III Motor test score-considered the benchmark for evaluating motor symptoms in individuals with PD-but also in various assessments such as the TUG test, TTT, and diverse gait features, as detailed in the White Papers on Proof of Concept from 2020. Moreover, users reported that donning the CUE1 device contributed to enhanced fatigue levels and increased subjective balance confidence.

Subsequent investigations from smaller-scale studies revealed notable advancements linked to CUE1 usage. Specifically, the device was shown to significantly boost gait speed in the TUG test (Tan et al., 2021) and improve MDS-UPDRS performance scores while reducing falls by an impressive 85% (Ong et al., 2022). Furthermore, a study design acceptance paper authored by Wilhelm et al. in 2022 showcased a reduction in Freezing of Gait (FOG) and an augmentation in walking speed, accompanied by positive feedback from individuals with PD regarding their experience with the CUE1.

This feasibility study will test primarily the feasibility, safety and tolerability and secondary the effect of the CUE1 and the CUE1+ (e.g., updated version of the CUE1 which has better motor and longer battery life but same treatment settings) device in people with PD and related disorders. This clinical study aims to identify whether the results seen in the prototype testing and previous small studies (Tan et al., 2021; Ong et al., 2022; Wilhelm et al., 2022) can be reproduced in a controlled clinical setting. Overall the risk assessment related to the use of the CUE1 and CUE1+ device has been previously tested on people with PD and has shown to have a minimal chance for error or adverse effect to the patient. Based on real world data, the CUE1 has shown to be effective in significantly improving motor symptoms such as rigidity, stiffness, tremor and slowness of movement in people with PD (White Paper-Proof of Concept, 2019; 2020). The CUE1 has also shown to improve fatigue (White Paper-Proof of Concept, 2020), walking speed, balance and FOG and decrease falls in people with PD (Tan et al., 2021; Ong et al., 2022; Wilhelm et al., 2022). The potential harm for the people with PD was very low, the acceptance of using the CUE1 and its renamed/rebranded model with longer battery life and better motor function, the CUE1+ device was very good, and positive user feedback was received (Wilhelm et al., 2022). The device also utilised medical grade established silicone-based skin adhesives. The product is water resistant and designed to CE standards hence product and electrical malfunction risk will be low.

Positive results arising from this feasibility study will strengthen the evidence that the CUE1+ device is feasible to be used, tolerated, safe and help to improve movement and mobility in people living with PD and related disorders. It may also assist in selecting the most appropriate outcome measures to test the effectiveness of the CUE1+ and contribute to the growing academic interest in the application of peripheral stimulation in other neurological disorders with movement, gait and balance problems such as various types of dystonias and tremors, multiple sclerosis, stroke and vestibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Clinical diagnosis of idiopathic PD and related disorders including progressive supranuclear palsy (PSP), multiple system atrophy (MSA), corticobasal degeneration (CBD), and vascular Parkinsonism (VaP) as well as atypical dystonias and tremor disorders and Orthostatic Tremor (OT)
* willing to participate and written consent provided after read the participant information sheet.

Exclusion Criteria:

Individuals with:

* other neurological disorders excluding idiopathic PD, related disorders such PSP, MSA, CBD, and VaP as well as atypical dystonias and tremor disorders, affecting movement, balance and gait
* metabolic or autoimmune disorders affecting movement, balance and gait
* acute orthopaedic disorders influencing balance control and gait
* audiovestibular disorders including severe hearing loss
* visual disturbances, poor eyesight
* not able to provide written consent form to participate
* clinical diagnosis of cognitive impairment including dementia or Alzheimer's.
* Mental impairments (illusions, hallucinations, impulse control disorders) (self-reported)

Technical contraindications related to CUE1 device:

* implanted metallic or electronic devices usage
* hypersensitivity to vibrotactile stimulation
* skin conditions and/or open wound in the area of where the device will be positioned (e.g., sternum) if taking medicines for PD or related disorder, then on stable dose of treatment for the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 minute
  This is a feasibility outcome, the recruitment rate which will be calculated as the percentage of eligible participants enrolled in the study. This will be reported at each follow up appointment at weeks -3, -6 and -9.
Compliance with interventions | 1 minute
  This is a feasibility outcome, compliance with interventions, which will be reported as the percentage of days completed using the CUE1 device and duration of using the CUE1 device. These will be reported at each follow up appointment at weeks -3, -6 and -9.
Dropout rate | 1 minute
  This is a feasibility outcome which will report the dropout rate at each follow up appointment at weeks -3, -6 and -9.
Physical observation | 1 minute
  This is a safety and tolerability outcome which will be assessed by carrying out a physical observation by research team during the face to face appointments of any adverse event occurring as a result of using the adhesive patches. The adverse events in relation to the CUE1 device will be reported in the participants' clinical diary and discussed during the appointments with the research team.

SECONDARY OUTCOMES:
Patient's Global Impression of Change (PGI-C) questionnaire | 5 minutes
  There are two parts in the PGI-C questionnaire. In part one, the patient scores on a scale 0-7 (0 = no change or condition has got worse, 7 = a great deal better, and a considerable improvement that has made all the difference) the change in their activity limitations, symptoms, emotions and overall QoL related to painful conditions. In part two, the patient scores on a scale 0-10 (0 = much better, 10 = much worse), the score that matches their degree of change since beginning the specific care (here the intervention with CUE1). The PGI-C will be completed at follow up appointments, at weeks-3, -6, and -9.
Participant's clinical diary | 15 minutes
  This will be completed daily by the participant at home for 9 weeks, starting from week-1 of and finishing at the end of week-9 of the intervention. The diaries will be completed on the weeks of the intervention (e.g., 1-2, 4-5 and 7-8). The research team will provide the same instructions on how to complete the participant's diary to each person during the baseline appointment at week-0.
Functional Gait Assessment (FGA) | 10 minutes
  The FGA is a 10-item test that assesses performance on complex gait tasks (i.e., walking with head turns, stepping over an obstacle, stopping and turning or climbing stairs). Scores for each item are between 0-3. The highest score is 30 and greater outcomes are indicative of better performance. The FGA has been validated in healthy people, older adults with a history of falls and balance impairments, and people with balance problems including those with PD. The minimal detectable change for the FGA is reported to be 4 points in people with PD. Scores ≤22/30 identify fall risk and are predictable of falls in community-living older persons within 6 months. In people with PD, the cutoff point for predicting falls is 18/30, with sensitivity of 80.6%, specificity of 80.0%, and positive likelihood ratio of 4.03.
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Motor Part III | 10 minutes
  The MDS-UPDRS Motor Part III assesses the motor symptoms in people with PD. There are 33 scores based on 18 questions with several right, left or other body distribution scores. All items have 5 response options with uniform anchors of 0 = normal, 1 = slight (symptoms/signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/signs of frequency or intensity sufficient to cause a modest impact on function), 3 = moderate (symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent function), and 4 = severe (symptoms/signs that prevent function). Higher scores indicate greater impact of PD symptoms. Score range between 0 and 132, 32 and below is mild, 59 and above is severe.
Timed Up and Go test (TUG) | 5 minutes
  The TUG assesses mobility, balance, walking ability, and fall risks. The mean time in people with PD has been reported between 10.3-14.8 seconds.
Bradykinesia Akinesia Incoordination test (BRAIN test) | 5 minutes
  The BRAIN test is used to assess upper limb motor function. The BRAIN test has been redeveloped to run in all internet browser software and has been validated in patients with PD and controls. Participants use the index finger of a single hand to alternately strike the 'S' and ';' keys on a standard computer keyboard, as fast and accurately as possible. The test is repeated for the other hand. The BRAIN test can be accessed at http://www.predictpd.com/braintest and applications to use this can be directed to AJN via the same web link.
Distal Finger Tapping (DFT) | 5 minutes
  The DFT test is a web-based keyboard tapping test which has been validated to remotely evaluate upper limb movements and quantify separate kinetic components such as speed, akinesia and rhythm as part of motor dysfunction in PD. It is available online via https://predictpd.com/en/braintest, and compatible with regular laptops and computers with a keyboard. The DFT test consists of a 20-second single key tapping test. Participants will be instructed to repeatedly tap the down arrow key with their left index finger, as fast as possible for 20 s, whilst simultaneously depressing the left arrow key with their left middle finger. The same task will then be repeated for the right hand. These instructions stabilise the wrist and forearm, isolating movement to the index finger metacarpal joint, thereby giving a true measurement of distal finger movement.
Activity-specific Balance Confidence (ABC) | 5 minutes
  The ABC is a 16-item questionnaire which assesses self-perceived balance confidence in daily activities. Scores range from 0-100; scores ≤ 67/100 are associated with increased fall risk. Higher scores indicate greater balance confidence.
Pittsburgh Sleep Quality Index (PSQI) | 5 minutes
  The PSQI includes seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medication, and daytime dysfunction. Scores range from 0-21 with a higher total score indicating worse sleep quality. In distinguishing good and poor sleepers, a global PSQI score > 5 yields sensitivity of 89.6% and specificity of 86.5%.
Fatigue Severity Scale (FSS) | 5 minutes
  The FSS is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders, including those with PD diagnosis. The items are scored on a 7-point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Parkinson's Disease Questionnaire (PDQ-39) | 5 minutes
  The PDQ-39 is a 39-item self-report questionnaire, which assesses PD-specific health related quality over the last month. It assesses how often patients experience difficulties across the 8 quality of life dimensions and impact of PD on specific dimensions of functioning and well-being. The scoring is done on a 5-point ordinal system (e.g., 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always). Each dimension's total score ranges from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (Parts I, II, IV). | 15 minutes
  The rest of the MDS-UPDRS scale consists of three parts (apart from Part III Motor which will be completed already above): Part I, II and IV which include questions to assess non-motor experiences of daily living, motor experiences of daily living, and motor complications, of people living with PD, respectively.
Participant's satisfaction form | 5 minutes
  This form will be will be provided to participants to complete at the last follow up appointment (week -9) to feedback on their experience on using the intervention, and support and services received from the research team.

OTHER OUTCOMES:
Age | within 1 minute
  Age is recorded in years and collected as baseline demographic characteristic only.
Gender | within 1 minute
  Gender is recorded as male, female, and other, and collected as baseline demographic characteristic only.
Disease duration | within 1 minute
  The disease duration is recorded in years and collected as baseline demographic characteristic only.
Hoehn & Yahr (H &Y) | within 1 minute
  Hoehn & Yahr (H & Y) scale is used to record the disease severity for people with Parkinson's disease.
Montreal Cognitive Assessment (MoCA) tool | within 5 minutes
  The MoCA is a rapid screening tool for mild cognitive impairment. It assesses different cognitive domains: attention and concentration, executive function, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. It has been recommended that cut-off scores of <26/30 be used to identify multi-domain cognitive impairment.
Cognitive Behavioural Symptom Questionnaire (CBSQ) | within 5 minutes
  The CBSQ is a measure of subjects' cognitive (i.e. beliefs) and behavioural responses to symptoms of their health condition. This measure includes five cognitive (i.e. beliefs) subscales: Symptom Focusing, Catastrophizing, Damaging Beliefs, Fear Avoidance and Embarrassment Avoidance; and two behavioural subscales: All or- Nothing and Avoidance/Rest. All items are rated on a 5-point Likert scale ranging from 'strongly disagree' to 'strongly agree'.
Illness Perception Questionnaire-Revised (IPQ-R) | within 5 minutes
  The IPQ-R was used to measure participants' illness perceptions. The IPQ-R measures the key components in Leventhal's common sense self-regulatory model: Illness identity was measured by asking patients to indicate whether they have experienced and attribute a number of potential symptoms to their dizziness condition, with higher scores (range 0-24) indicating increased illness identity. In accordance with the recommendations from the authors, some items were added based on feedback from a patient-public involvement group so as to reflect the symptoms experienced by people with vestibular disorders. Causal Factors were measured by asking participants to list up to three things that they believed caused their condition.
Falls questionnaire | within 15 minutes
  This has four main sections: a) Symptom Severity; b) Symptom Frequency; c) Balance and Falls: Details on balance, gait, falls, costs, care received, and the impact on QoL, rated on a 0-10 scale; d) Standard Care: Information on type, frequency, duration, perceived benefit, and adverse reactions. Group A also includes a fifth section on the CUE1, covering open- and closed-ended questions on usability, safety, tolerability, and its effects on symptoms, independence, QoL, mood, social interaction, fear of falling, and balance confidence.
Parkinson's KinetiGraph | every day for the duration of the study, 24 h a day
  Parkinson's KinetiGraph (PKG) (Odin et al. 2018) is a wrist worn logger-watch developed by the Global Kinetics Pty Ltd. Accelerometry data is recorded by the PKG watch while worn on wrist for the duration of the study starting from the baseline appointment and finishing at the 3 month follow up appointment. Participants will be wearing the PKG watch at all times while they continue their regular activities of daily living and taking it off only when they need to charge it.
Ethnicity | less than 1 minute
  White or White British (n, %) Mixed or multiple ethnic group (n, %) Asian or Asian British (n, %) Black, African, Caribbean or Black British Another ethnic group

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Noyce, PhD, Study Director — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

REFERENCES:
- [Background] Akram N, Li H, Ben-Joseph A, Budu C, Gallagher DA, Bestwick JP, Schrag A, Noyce AJ, Simonet C. Developing and assessing a new web-based tapping test for measuring distal movement in Parkinson's disease: a Distal Finger Tapping test. Sci Rep. 2022 Jan 10;12(1):386. doi: 10.1038/s41598-021-03563-7. PMID 35013372
- [Background] Basta D, Rossi-Izquierdo M, Soto-Varela A, Greters ME, Bittar RS, Steinhagen-Thiessen E, Eckardt R, Harada T, Goto F, Ogawa K, Ernst A. Efficacy of a vibrotactile neurofeedback training in stance and gait conditions for the treatment of balance deficits: a double-blind, placebo-controlled multicenter study. Otol Neurotol. 2011 Dec;32(9):1492-9. doi: 10.1097/MAO.0b013e31823827ec. PMID 22089958
- [Background] Beck EN, Ehgoetz Martens KA, Almeida QJ. Freezing of Gait in Parkinson's Disease: An Overload Problem? PLoS One. 2015 Dec 17;10(12):e0144986. doi: 10.1371/journal.pone.0144986. eCollection 2015. PMID 26678262
- [Background] Bloem BR, Grimbergen YA, Cramer M, Valkenburg VV. "Stops walking when talking" does not predict falls in Parkinson's disease. Ann Neurol. 2000 Aug;48(2):268. doi: 10.1002/1531-8249(200008)48:23.0.co;2-4. No abstract available. PMID 10939582
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chaudhuri KR, Schrag A, Weintraub D, Rizos A, Rodriguez-Blazquez C, Mamikonyan E, Martinez-Martin P. The movement disorder society nonmotor rating scale: Initial validation study. Mov Disord. 2020 Jan;35(1):116-133. doi: 10.1002/mds.27862. Epub 2019 Sep 30. PMID 31571279
- [Background] Chomiak T, Watts A, Meyer N, Pereira FV, Hu B. A training approach to improve stepping automaticity while dual-tasking in Parkinson's disease: A prospective pilot study. Medicine (Baltimore). 2017 Feb;96(5):e5934. doi: 10.1097/MD.0000000000005934. PMID 28151878
- [Background] Conte A, Khan N, Defazio G, Rothwell JC, Berardelli A. Pathophysiology of somatosensory abnormalities in Parkinson disease. Nat Rev Neurol. 2013 Dec;9(12):687-97. doi: 10.1038/nrneurol.2013.224. Epub 2013 Nov 12. PMID 24217516
- [Background] Dal Bello-Haas V, Klassen L, Sheppard MS, Metcalfe A. Psychometric Properties of Activity, Self-Efficacy, and Quality-of-Life Measures in Individuals with Parkinson Disease. Physiother Can. 2011 Winter;63(1):47-57. doi: 10.3138/ptc.2009-08. Epub 2011 Jan 20. PMID 22210979
- [Background] Dincher A, Schwarz M, Wydra G. Analysis of the Effects of Whole-Body Vibration in Parkinson Disease - Systematic Review and Meta-Analysis. PM R. 2019 Jun;11(6):640-653. doi: 10.1002/pmrj.12094. Epub 2019 May 6. PMID 30689308
- [Background] Dorsey ER, Sherer T, Okun MS, Bloem BR. The Emerging Evidence of the Parkinson Pandemic. J Parkinsons Dis. 2018;8(s1):S3-S8. doi: 10.3233/JPD-181474. PMID 30584159
- [Background] Farombi TH, Owolabi MO, Ogunniyi A. Falls and Their Associated Risks in Parkinson's Disease Patients in Nigeria. J Mov Disord. 2016 Sep;9(3):160-5. doi: 10.14802/jmd.16011. Epub 2016 Sep 21. PMID 27667188
- [Background] Fok P, Farrell M, McMeeken J. Prioritizing gait in dual-task conditions in people with Parkinson's. Hum Mov Sci. 2010 Oct;29(5):831-42. doi: 10.1016/j.humov.2010.06.005. Epub 2010 Aug 19. PMID 20727609
- [Background] Giladi N, Shabtai H, Simon ES, Biran S, Tal J, Korczyn AD. Construction of freezing of gait questionnaire for patients with Parkinsonism. Parkinsonism Relat Disord. 2000 Jul 1;6(3):165-170. doi: 10.1016/s1353-8020(99)00062-0. PMID 10817956
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Goncalves H, Moreira R, Rodrigues A, Santos C. Finding Parameters around the Abdomen for a Vibrotactile System: Healthy and Patients with Parkinson's Disease. J Med Syst. 2018 Oct 13;42(11):232. doi: 10.1007/s10916-018-1087-2. PMID 30317396
- [Background] Grosset D, Taurah L, Burn DJ, MacMahon D, Forbes A, Turner K, Bowron A, Walker R, Findley L, Foster O, Patel K, Clough C, Castleton B, Smith S, Carey G, Murphy T, Hill J, Brechany U, McGee P, Reading S, Brand G, Kelly L, Breen K, Ford S, Baker M, Williams A, Hearne J, Qizilbash N, Chaudhuri KR. A multicentre longitudinal observational study of changes in self reported health status in people with Parkinson's disease left untreated at diagnosis. J Neurol Neurosurg Psychiatry. 2007 May;78(5):465-9. doi: 10.1136/jnnp.2006.098327. Epub 2006 Nov 10. PMID 17098846
- [Background] Hasan H, Burrows M, Athauda DS, Hellman B, James B, Warner T, Foltynie T, Giovannoni G, Lees AJ, Noyce AJ. The BRadykinesia Akinesia INcoordination (BRAIN) Tap Test: Capturing the Sequence Effect. Mov Disord Clin Pract. 2019 Jun 25;6(6):462-469. doi: 10.1002/mdc3.12798. eCollection 2019 Jul. PMID 31392247
- [Background] Heremans E, Nackaerts E, Vervoort G, Broeder S, Swinnen SP, Nieuwboer A. Impaired Retention of Motor Learning of Writing Skills in Patients with Parkinson's Disease with Freezing of Gait. PLoS One. 2016 Feb 10;11(2):e0148933. doi: 10.1371/journal.pone.0148933. eCollection 2016. PMID 26862915
- [Background] Hoops S, Nazem S, Siderowf AD, Duda JE, Xie SX, Stern MB, Weintraub D. Validity of the MoCA and MMSE in the detection of MCI and dementia in Parkinson disease. Neurology. 2009 Nov 24;73(21):1738-45. doi: 10.1212/WNL.0b013e3181c34b47. PMID 19933974
- [Background] Huber M, Knottnerus JA, Green L, van der Horst H, Jadad AR, Kromhout D, Leonard B, Lorig K, Loureiro MI, van der Meer JW, Schnabel P, Smith R, van Weel C, Smid H. How should we define health? BMJ. 2011 Jul 26;343:d4163. doi: 10.1136/bmj.d4163. No abstract available. PMID 21791490
- [Background] Hurst H, Bolton J. Assessing the clinical significance of change scores recorded on subjective outcome measures. J Manipulative Physiol Ther. 2004 Jan;27(1):26-35. doi: 10.1016/j.jmpt.2003.11.003. PMID 14739871
- [Background] Isaacson S, O'Brien A, Lazaro JD, Ray A, Fluet G. The JFK BIG study: the impact of LSVT BIG(R) on dual task walking and mobility in persons with Parkinson's disease. J Phys Ther Sci. 2018 Apr;30(4):636-641. doi: 10.1589/jpts.30.636. Epub 2018 Apr 20. PMID 29706722
- [Background] Jacobs JV, Nutt JG, Carlson-Kuhta P, Allen R, Horak FB. Dual tasking during postural stepping responses increases falls but not freezing in people with Parkinson's disease. Parkinsonism Relat Disord. 2014 Jul;20(7):779-81. doi: 10.1016/j.parkreldis.2014.04.001. Epub 2014 Apr 14. PMID 24768615
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Killane I, Fearon C, Newman L, McDonnell C, Waechter SM, Sons K, Lynch T, Reilly RB. Dual Motor-Cognitive Virtual Reality Training Impacts Dual-Task Performance in Freezing of Gait. IEEE J Biomed Health Inform. 2015 Nov;19(6):1855-61. doi: 10.1109/JBHI.2015.2479625. Epub 2015 Sep 17. PMID 26394439
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Lajoie Y, Gallagher SP. Predicting falls within the elderly community: comparison of postural sway, reaction time, the Berg balance scale and the Activities-specific Balance Confidence (ABC) scale for comparing fallers and non-fallers. Arch Gerontol Geriatr. 2004 Jan-Feb;38(1):11-26. doi: 10.1016/s0167-4943(03)00082-7. PMID 14599700
- [Background] Lamont RM, Morris ME, Menz HB, McGinley JL, Brauer SG. Falls in people with Parkinson's disease: A prospective comparison of community and home-based falls. Gait Posture. 2017 Jun;55:62-67. doi: 10.1016/j.gaitpost.2017.04.005. Epub 2017 Apr 4. PMID 28419875
- [Background] Leddy AL, Crowner BE, Earhart GM. Functional gait assessment and balance evaluation system test: reliability, validity, sensitivity, and specificity for identifying individuals with Parkinson disease who fall. Phys Ther. 2011 Jan;91(1):102-13. doi: 10.2522/ptj.20100113. Epub 2010 Nov 11. PMID 21071506
- [Background] Mak MK, Yu L, Hui-Chan CW. The immediate effect of a novel audio-visual cueing strategy (simulated traffic lights) on dual-task walking in people with Parkinson's disease. Eur J Phys Rehabil Med. 2013 Apr;49(2):153-9. Epub 2013 Mar 13. PMID 23480976
- [Background] Mancini M, Smulders K, Harker G, Stuart S, Nutt JG. Assessment of the ability of open- and closed-loop cueing to improve turning and freezing in people with Parkinson's disease. Sci Rep. 2018 Aug 24;8(1):12773. doi: 10.1038/s41598-018-31156-4. PMID 30143726
- [Background] Marchetti GF, Lin CC, Alghadir A, Whitney SL. Responsiveness and minimal detectable change of the dynamic gait index and functional gait index in persons with balance and vestibular disorders. J Neurol Phys Ther. 2014 Apr;38(2):119-24. doi: 10.1097/NPT.0000000000000015. PMID 24637931
- [Background] Muthukrishnan N, Abbas JJ, Shill HA, Krishnamurthi N. Cueing Paradigms to Improve Gait and Posture in Parkinson's Disease: A Narrative Review. Sensors (Basel). 2019 Dec 11;19(24):5468. doi: 10.3390/s19245468. PMID 31835870
- [Background] Muslimovic D, Post B, Speelman JD, Schmand B, de Haan RJ; CARPA Study Group. Determinants of disability and quality of life in mild to moderate Parkinson disease. Neurology. 2008 Jun 3;70(23):2241-7. doi: 10.1212/01.wnl.0000313835.33830.80. PMID 18519873
- [Background] Munoz-Hellin E, Cano-de-la-Cuerda R, Miangolarra-Page JC. [Visual cues as a therapeutic tool in Parkinson's disease. A systematic review]. Rev Esp Geriatr Gerontol. 2013 Jul-Aug;48(4):190-7. doi: 10.1016/j.regg.2013.03.002. Epub 2013 Jun 2. Spanish. PMID 23735596
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Nieuwboer A, Kwakkel G, Rochester L, Jones D, van Wegen E, Willems AM, Chavret F, Hetherington V, Baker K, Lim I. Cueing training in the home improves gait-related mobility in Parkinson's disease: the RESCUE trial. J Neurol Neurosurg Psychiatry. 2007 Feb;78(2):134-40. doi: 10.1136/jnnp.200X.097923. PMID 17229744
- [Background] Noyce AJ, Nagy A, Acharya S, Hadavi S, Bestwick JP, Fearnley J, Lees AJ, Giovannoni G. Bradykinesia-akinesia incoordination test: validating an online keyboard test of upper limb function. PLoS One. 2014 Apr 29;9(4):e96260. doi: 10.1371/journal.pone.0096260. eCollection 2014. PMID 24781810
- [Background] Nutt JG, Bloem BR, Giladi N, Hallett M, Horak FB, Nieuwboer A. Freezing of gait: moving forward on a mysterious clinical phenomenon. Lancet Neurol. 2011 Aug;10(8):734-44. doi: 10.1016/S1474-4422(11)70143-0. PMID 21777828
- [Background] Otis MJ, Ayena JC, Tremblay LE, Fortin PE, Menelas BA. Use of an Enactive Insole for Reducing the Risk of Falling on Different Types of Soil Using Vibrotactile Cueing for the Elderly. PLoS One. 2016 Sep 7;11(9):e0162107. doi: 10.1371/journal.pone.0162107. eCollection 2016. PMID 27603211
- [Background] Park JK, Kim SJ. Dual-Task-Based Drum Playing with Rhythmic Cueing on Motor and Attention Control in Patients with Parkinson's Disease: A Preliminary Randomized Study. Int J Environ Res Public Health. 2021 Sep 26;18(19):10095. doi: 10.3390/ijerph181910095. PMID 34639396
- [Background] Pereira MP, Gobbi LT, Almeida QJ. Freezing of gait in Parkinson's disease: Evidence of sensory rather than attentional mechanisms through muscle vibration. Parkinsonism Relat Disord. 2016 Aug;29:78-82. doi: 10.1016/j.parkreldis.2016.05.021. Epub 2016 May 21. PMID 27245918
- [Background] Pfeifer KJ, Kromer JA, Cook AJ, Hornbeck T, Lim EA, Mortimer BJP, Fogarty AS, Han SS, Dhall R, Halpern CH, Tass PA. Coordinated Reset Vibrotactile Stimulation Induces Sustained Cumulative Benefits in Parkinson's Disease. Front Physiol. 2021 Apr 6;12:624317. doi: 10.3389/fphys.2021.624317. eCollection 2021. PMID 33889086
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Redgrave P, Rodriguez M, Smith Y, Rodriguez-Oroz MC, Lehericy S, Bergman H, Agid Y, DeLong MR, Obeso JA. Goal-directed and habitual control in the basal ganglia: implications for Parkinson's disease. Nat Rev Neurosci. 2010 Nov;11(11):760-72. doi: 10.1038/nrn2915. Epub 2010 Oct 14. PMID 20944662
- [Background] Rochester L, Baker K, Hetherington V, Jones D, Willems AM, Kwakkel G, Van Wegen E, Lim I, Nieuwboer A. Evidence for motor learning in Parkinson's disease: acquisition, automaticity and retention of cued gait performance after training with external rhythmical cues. Brain Res. 2010 Mar 10;1319:103-11. doi: 10.1016/j.brainres.2010.01.001. Epub 2010 Jan 11. PMID 20064492
- [Background] Rochester L, Burn DJ, Woods G, Godwin J, Nieuwboer A. Does auditory rhythmical cueing improve gait in people with Parkinson's disease and cognitive impairment? A feasibility study. Mov Disord. 2009 Apr 30;24(6):839-45. doi: 10.1002/mds.22400. PMID 19199354
- [Background] Rochester L, Nieuwboer A, Baker K, Hetherington V, Willems AM, Chavret F, Kwakkel G, Van Wegen E, Lim I, Jones D. The attentional cost of external rhythmical cues and their impact on gait in Parkinson's disease: effect of cue modality and task complexity. J Neural Transm (Vienna). 2007;114(10):1243-8. doi: 10.1007/s00702-007-0756-y. Epub 2007 Jun 28. PMID 17598068
- [Background] Rochester L, Rafferty D, Dotchin C, Msuya O, Minde V, Walker RW. The effect of cueing therapy on single and dual-task gait in a drug naive population of people with Parkinson's disease in northern Tanzania. Mov Disord. 2010 May 15;25(7):906-11. doi: 10.1002/mds.22978. PMID 20175212
- [Background] Tan XS, Pierres F, Dallman-Porter A, Hardie-Brown W, Kwon KY. Focused Vibrotactile Stimulation with Cueing Effect on Freezing of Gait in Parkinson's Disease: Two Case Reports. J Mov Disord. 2021 Sep;14(3):236-238. doi: 10.14802/jmd.21076. Epub 2021 Sep 8. PMID 34488302
- [Background] Shribman S, Hasan H, Hadavi S, Giovannoni G, Noyce AJ. The BRAIN test: a keyboard-tapping test to assess disability and clinical features of multiple sclerosis. J Neurol. 2018 Feb;265(2):285-290. doi: 10.1007/s00415-017-8690-x. Epub 2017 Dec 4. PMID 29204963
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Skerrett TN, Moss-Morris R. Fatigue and social impairment in multiple sclerosis: the role of patients' cognitive and behavioral responses to their symptoms. J Psychosom Res. 2006 Nov;61(5):587-93. doi: 10.1016/j.jpsychores.2006.04.018. PMID 17084135
- [Background] Spaulding SJ, Barber B, Colby M, Cormack B, Mick T, Jenkins ME. Cueing and gait improvement among people with Parkinson's disease: a meta-analysis. Arch Phys Med Rehabil. 2013 Mar;94(3):562-70. doi: 10.1016/j.apmr.2012.10.026. Epub 2012 Nov 2. PMID 23127307
- [Background] Stuart S, Mancini M. Prefrontal Cortical Activation With Open and Closed-Loop Tactile Cueing When Walking and Turning in Parkinson Disease: A Pilot Study. J Neurol Phys Ther. 2020 Apr;44(2):121-131. doi: 10.1097/NPT.0000000000000286. PMID 31425309
- [Background] van Wegen E, de Goede C, Lim I, Rietberg M, Nieuwboer A, Willems A, Jones D, Rochester L, Hetherington V, Berendse H, Zijlmans J, Wolters E, Kwakkel G. The effect of rhythmic somatosensory cueing on gait in patients with Parkinson's disease. J Neurol Sci. 2006 Oct 25;248(1-2):210-4. doi: 10.1016/j.jns.2006.05.034. Epub 2006 Jun 14. PMID 16780887
- [Background] Volpe D, Giantin MG, Fasano A. A wearable proprioceptive stabilizer (Equistasi(R)) for rehabilitation of postural instability in Parkinson's disease: a phase II randomized double-blind, double-dummy, controlled study. PLoS One. 2014 Nov 17;9(11):e112065. doi: 10.1371/journal.pone.0112065. eCollection 2014. PMID 25401967
- [Background] Wagle Shukla A, Ounpraseuth S, Okun MS, Gray V, Schwankhaus J, Metzer WS. Micrographia and related deficits in Parkinson's disease: a cross-sectional study. BMJ Open. 2012 Jun 25;2(3):e000628. doi: 10.1136/bmjopen-2011-000628. Print 2012. PMID 22734114
- [Background] Weir S, Samnaliev M, Kuo TC, Tierney TS, Walleser Autiero S, Taylor RS, Schrag A. Short- and long-term cost and utilization of health care resources in Parkinson's disease in the UK. Mov Disord. 2018 Jul;33(6):974-981. doi: 10.1002/mds.27302. Epub 2018 Mar 30. PMID 29603405
- [Background] Wilhelm A, Riedl T, Paumann C, Janssen J. Exploring a New Cueing Device in People Who Experience Freezing of Gait: Acceptance of a Study Design. Parkinsons Dis. 2022 Dec 7;2022:1631169. doi: 10.1155/2022/1631169. eCollection 2022. PMID 37250383
- [Background] Wrisley DM, Kumar NA. Functional gait assessment: concurrent, discriminative, and predictive validity in community-dwelling older adults. Phys Ther. 2010 May;90(5):761-73. doi: 10.2522/ptj.20090069. Epub 2010 Apr 1. PMID 20360052
- [Background] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- [Background] Yang Y, Wang Y, Zhou Y, Chen C, Xing D, Wang C. Validity of the Functional Gait Assessment in patients with Parkinson disease: construct, concurrent, and predictive validity. Phys Ther. 2014 Mar;94(3):392-400. doi: 10.2522/ptj.20130019. Epub 2013 Oct 24. PMID 24158644
- [Background] Yang Y, Wang Y, Zhou Y, Chen C, Xing D. Reliability of functional gait assessment in patients with Parkinson disease: Interrater and intrarater reliability and internal consistency. Medicine (Baltimore). 2016 Aug;95(34):e4545. doi: 10.1097/MD.0000000000004545. PMID 27559954
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Derived] Azoidou V, Bhadra E, Rowsell K, Camboe E, Dey K, Zirra A, Quah C, Budu C, Boyle T, Gallagher D, Noyce A, Simonet C. Non-invasive device to alleviate symptoms in people living with Parkinson's: study protocol for a multicentre phase II double-blind randomised controlled trial. BMJ Open. 2025 Apr 27;15(4):e096051. doi: 10.1136/bmjopen-2024-096051. PMID 40288787
- See also: A Pilot Interventional Study on Feasibility and Effectiveness of the CUE1 device in Parkinson's disease-first results in manuscript — https://doi.org/10.1101/2024.10.11.24315305